CLINICAL TRIAL: NCT06350591
Title: Evaluating Changes in Skeletal Muscle Protein Synthesis, and the Dynamic Proteome, Following Unilateral Resistance Exercise Training and Single-leg Immobilization
Brief Title: Evaluating Changes in Skeletal Muscle Proteins Following Resistance Exercise and Single-Leg Disuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Chris McGlory, PhD, Assistant Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6038674
Record Dates: First submitted 2024-01-16; First posted 2024-04-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Skeletal Muscle Atrophy; Skeletal Muscle Hypertrophy
MeSH Terms: conditions — Muscular Atrophy | interventions — Immobilization; Resistance Training

STUDY DESIGN:
Intervention Model Description: parallel, within-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immobilization (Experimental): Participants will undergo 10 days of unilateral immobilization whereby a leg will remain in 60 degrees of flexion with the use of a brace. All participants will complete this protocol.
  Interventions: Other: Immobilization
- Resistance Training (Experimental): Participants will undergo 4 sessions of unilateral resistance training over a 10 day period (the resistance training protocol will include 3 sets of 8-12 reps of leg press and leg extension). All participants will complete this protocol. On day 0, participants will be asked to undergo a bout of unilateral resistance exercise, and the investigators will assess the acute response to exercise + protein feeding (via EAA supplement).
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Immobilization — single-leg immobilization
  Arms: Immobilization
Other: Resistance training — Leg extension and leg press; 3 sets of 8-12 reps
  Arms: Resistance Training

SUMMARY:
Skeletal muscle plays a critical role in supporting human health. Beyond its role in providing the force to move, skeletal muscle accounts for a large proportion of metabolic rate, glucose disposal, and amino acid storage. Skeletal muscle is dynamically regulated by environmental stimuli, such as loading (i.e., resistance training]) and unloading (i.e., disuse atrophy) as well as the intake of essential amino acids (EAAs). However, the precise mechanisms that regulate skeletal muscle mass in response to various conditions (e.g., EAA supplementation, resistance training, and unloading) are not completely understood. Therefore, concerted efforts to better understand the mechanisms regulating skeletal muscle size are needed that aid in the development of therapeutic interventions to combat age, disease, and disuse related muscular atrophy.

DETAILED DESCRIPTION:
Skeletal muscle is a highly plastic tissue capable of modifying its phenotype (i.e., structural, contractile, and metabolic properties) in response to alterations in mechanical loading. Mechanistically underpinning skeletal muscle plasticity are changes in skeletal muscle protein turnover. Skeletal muscle size is dictated by changes in rates of muscle protein synthesis (MPS) and rates of muscle protein breakdown (MPB) with changes in rates of MPS being the primary determinant of human skeletal muscle mass. Both MPS and MPB are highly sensitive to contractile and nutritional cues. In response to EAA ingestion, there is a rise in rates of MPS and a mild suppression of MPB rates resulting in a positive state of protein balance. Similarly, when an individual performs a bout of resistance exercise, there is an increase in rates of MPS that is potentiated by EAA feeding; It is for this reason that when repeated bouts of resistance exercise are coupled with EAA intake over time, there is a gradual increase in skeletal muscle mass termed hypertrophy. In contrast, when an individual undergoes a reduction in levels of contractile activity (e.g., immobilization due to injury or surgery), there is a reduction in both fed and fasted rates of MPS leading to the loss of skeletal muscle mass and size termed muscle atrophy.

Although it is well known that both nutrition and contractile activity affect rates of muscle protein turnover and skeletal muscle mass, our current knowledge is limited by most studies reporting rates of MPS and MPB that are averages of thousands of proteins in the whole muscle, or subcellular protein fractions, such as myofibrillar, sarcoplasmic, and mitochondrial. Further, individual protein MPS and MPB rates might span a broad range and there may be selective changes to the turnover of individual proteins under different skeletal muscle loading scenarios. Dynamic proteomic profiling (DPP) is an emerging methodology that combines quantitative proteomic abundance measurements with individual protein MPS and MPB rates, to deliver unprecedented insight into the molecular regulation of individual protein turnover. Another major consideration is that nearly all studies in this field have been conducted in males, with limited data in females. The lack of data in females is a major knowledge gap and of major concern particularly given there is evidence that women may display different molecular responses to exercise, nutrition, and disuse compared to men.

The purpose of this investigation is to gain a better understanding of the acute and short-term effects of an EAA supplement and an acute bout of resistance exercise on rates of muscle protein turnover. Further, the investigators aim to measure the dynamic proteome during 10 days of unilateral leg immobilization, and following several bouts of resistance exercise in the contralateral leg, in young healthy women. The present investigation will characterize skeletal muscle mass, strength, protein expression, and protein synthesis rates (individual [i.e., DPP] and average). The study may inform potential future novel interventions to attenuate losses in skeletal muscle mass owing to disuse, aging, or injury.

ELIGIBILITY:
Inclusion Criteria:

* Females 18-30 years
* BMI between 18-28 kg/m2
* ≥2 days per week of structured exercise
* Generally healthy as assessed by medical and physical activity questionnaires
* Participants not currently pregnant

Exclusion Criteria:

* Any muscular, neurological, respiratory, or metabolic disease including diabetes
* Any form of cancer currently or in the last 5 years
* Bleeding disorders or antiplatelet / anticoagulation therapy
* Currently taking fish oils or within the last 6 months
* Currently taking any form of steroid or within the last 3 months
* Inability to attain magnetic resonance imaging scans
* Known irregular responses to physical activity (e.g., shortness of breath, chest pain, dizziness, etc.)
* Any current illness
* Currently smoking or smoking within the last 6 months
* Currently pregnant
* Any concurrent medical, psychiatric, or orthopedic condition that, subject to investigators' discernment, would negatively affect the subject's ability to comply with the study requirements

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in average rates of muscle synthesis | -2, 0 (-4, 0, and 4 hours), and 10 days
  Skeletal muscle amino acids will be isolated and derivatized. Deuterium enrichment into protein-bound alanine will be measured using Gas chromatography-Pyrolysis-Isotope Ratio Mass Spectrometry
Dynamic proteomic profiling | -2, 0, and 10 days
  Skeletal muscle lysates containing ~100 ug protein will be digested using sequencing-grade trypsin, and analyzed, via UPLC-QTOF-MS. This will enable the quantification of changes in individual protein abundance, and rates of synthesis and breakdown.

SECONDARY OUTCOMES:
Protein expression (phosphorylation and content) of novel and known targets implicated in protein translation and mitochondrial-related protein expression | 0 (-4, 0, and 4 hours), and 10 days
  Translational factors and novel proteins involved in skeletal muscle protein synthesis (e.g. mTORC1, p70S6K1, Deptor, NID2, FKBP1A, BCAT2, MBNL1, AGO2, LRRC30, and TP53BP1), and mitochondrial function (e.g., ANT1) will be assessed, via western blotting
Muscle torque | -6 and 10 days
  Muscle torque will be measured during seated isometric knee extension on a dynamometer
Quadriceps skeletal muscle volume | 0 and 10 days
  Quadriceps muscle volume assessed by magnetic resonance imaging scan.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Kinesiology and Health Studies, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No